CLINICAL TRIAL: NCT02939820
Title: Expanded Access Protocol of Patisiran for Patients With Hereditary Transthyretin-Mediated Amyloidosis (hATTR Amyloidosis) With Polyneuropathy
Brief Title: Expanded Access Protocol of Patisiran for Patients With Hereditary ATTR Amyloidosis (hATTR)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-TTR02-007
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: TTR-mediated Amyloidosis; Amyloidosis, Hereditary; Amyloid Neuropathies, Familial; Familial Amyloid Polyneuropathies; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related
Keywords: RNAi therapeutic; FAP; Familial Amyloid Polyneuropathies; TTR; Transthyretin; Amyloidosis
MeSH Terms: conditions — Amyloidosis, Familial; Amyloid Neuropathies, Familial; Amyloid Neuropathies; Amyloidosis, Hereditary, Transthyretin-Related; Amyloidosis | interventions — patisiran

INTERVENTIONS:
Drug: patisiran (ALN-TTR02) — patisiran (ALN-TTR02) administered by intravenous (IV) infusion

SUMMARY:
The purpose of this study is to provide expanded access of patisiran to patients with hereditary transthyretin-mediated amyloidosis (hATTR).

DETAILED DESCRIPTION:
Choosing to participate in an expanded access program is an important personal decision. Talk with your doctor and family members or friends about deciding to join a research study. To learn more about this study, please have your doctor contact the study research staff using the Contacts provided. For general information, see the links provided in More Information.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than or equal to 18 years of age
* Have a diagnosis of hATTR
* Meet Karnofsky performance status and Polyneuropathy Disability (PND) score requirements
* Have adequate complete blood counts, liver function tests and coagulation tests

Exclusion Criteria:

* Participated in an interventional hATTR amyloidosis clinical trial involving RNA interference (RNAi) therapeutics within the last 12 months
* Are currently eligible to participate in or currently enrolled in an ongoing interventional hATTR amyloidosis clinical trial
* Have inadequate cardiac function
* Known primary amyloidosis (AL amyloidosis) or leptomeningeal amyloidosis
* Have known serious comorbidities or considered unfit for the program by the investigator
* Prior or planned liver or heart transplantation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals

REFERENCES:
- [Derived] Miah KM, Hyde SC, Gill DR. Emerging gene therapies for cystic fibrosis. Expert Rev Respir Med. 2019 Aug;13(8):709-725. doi: 10.1080/17476348.2019.1634547. Epub 2019 Jun 27. PMID 31215818
- See also: https://ghr.nlm.nih.gov/condition/transthyretin-amyloidosis — https://ghr.nlm.nih.gov/condition/transthyretin-amyloidosis
- See also: https://www.nlm.nih.gov/medlineplus/amyloidosis.html — https://www.nlm.nih.gov/medlineplus/amyloidosis.html